CLINICAL TRIAL: NCT01668823
Title: A Phase I Study of Light Dose for Photodynamic Therapy(PDT) Using 2-[ 1-hexyloxyethel]-2-devinyl Pyropheophorbide-a (HPPH) for Treatment of Non-small Cell Carcinoma in Situ or Non-small Cell Microinvasive Carcinoma. A Dose Ranging Study
Brief Title: Photodynamic Therapy in Treating Patients With Lung Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: I 05903; NCI-2010-02114 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2012-08-16; First posted 2012-08-20 (Estimated); Last update posted 2014-07-31 (Estimated); Status verified 2014-07

CONDITIONS: Adenocarcinoma of the Lung; Large Cell Lung Cancer; Recurrent Non-small Cell Lung Cancer; Squamous Cell Lung Cancer; Stage 0 Non-small Cell Lung Cancer
MeSH Terms: conditions — Adenocarcinoma of Lung; Carcinoma, Non-Small-Cell Lung | interventions — 2-(1-hexyloxyethyl)-2-devinyl pyropheophorbide-a; Photochemotherapy; 1-phenyl-3,3-dimethyltriazene

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (PDT using HPPH) (Experimental): Patients receive HPPH IV over 1 hour on day 1. Patients then photodynamic therapy with laser light on day 3. Patients also undergo therapeutic bronchoscopy for endoscopic debridement on day 5.
  Interventions: Drug: HPPH; Drug: photodynamic therapy; Procedure: therapeutic bronchoscopy

INTERVENTIONS:
Drug: HPPH — Given IV
  Other Names: Photochlor
Drug: photodynamic therapy — Undergo photodynamic therapy with HPPH
  Other Names: Light Infusion Therapy™; PDT; therapy, photodynamic
Procedure: therapeutic bronchoscopy — Undergo therapeutic bronchoscopy for endoscopic debridement

SUMMARY:
This phase I trial is studying the side effects and best dose of photodynamic therapy using HPPH in treating patients with lung cancer. Photodynamic therapy uses a drug, such as HPPH, that becomes active when it is exposed to a certain kind of light. When the drug is active, cancer cells are killed.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine maximally tolerated light dose (MTID). Identify systemic and normal tissue toxicity using 2-[hexyloxyethyl)-2-devinyl pyropheophorbide-a (HPPH) for photodynamic therapy in patients with bronchogenic carcinoma-in-situ (CIS) or microinvasive carcinoma.

SECONDARY OBJECTIVES:

I. To study tumor response in patients with bronchogenic carcinoma-in-situ (CIS) or bronchogenic microinvasive carcinoma.

OUTLINE: This is a dose-escalation study.

Patients receive HPPH intravenously (IV) over 1 hour on day 1. Patients then photodynamic therapy with laser light on day 3. Patients also undergo therapeutic bronchoscopy for endoscopic debridement on day 5.

After completion of study treatment, patients are followed up at 4-6 weeks, 6 months, and then periodically for at least 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients with biopsy confirmed carcinoma-in-situ (CIS) or microinvasive lung cancer
* Patients may have squamous cell carcinoma, adenocarcinoma, or large cell carcinoma
* Patients may have received prior therapy for lung cancer of any type, e.g. chemotherapy, radiation therapy
* Patients must have no contraindications for bronchoscopy
* Female patients must not be pregnant and must be practicing a medically acceptable form of birth control, be sterile or post-menopausal
* Patients must have a Karnofsky scale 50 or above (Eastern Cooperative Oncology Group [ECOG] 0-2)
* Patients must sign an Informed Consent according to Food and Drug Administration (FDA) guidelines acceptable to the Roswell Park Cancer Institute (RPCI) Institutional Review Board (IRB)
* Patients with underlying lung disease must be judged (by the principal investigator) able to with stand mucous/debris formation at the site of treatment
* Definition of CIS or microinvasive lung cancer for this protocol: the lesion will be radiographically occult and not definable by conventional computed tomography (CT) of the chest; the lesion may or may not be invisible on white light bronchoscopy, but is definable and photographable on lung imaging fluorescence endoscope (LIFE) bronchoscopy; biopsies of the lesion must indicate no evidence of invasion beyond cartilage on histopathology; the lesion may, however, be invasive through the basement membrane (microinvasive carcinoma)

Exclusion Criteria:

* Porphyria or hypersensitivity to porphyrin or porphyrin-like compounds
* White blood cells (WBC) < 4000
* Platelet count < 100,000
* Prothrombin time exceeding 1.5 times the upper normal limit
* Total serum bilirubin > 3.0 mg/dl
* Serum creatinine > 3.0 mg/dl
* Alkaline phosphatase (hepatic) or serum glutamic oxaloacetic transaminase (SGOT) > 3 times the upper normal limit
* Severe chronic obstructive pulmonary disease (COPD) that would in the opinion of the investigator preclude multiple bronchoscopies or partial central airway obstruction from mucous/debris formation
* Any evidence of worsening pulmonary symptoms or COPD exacerbation
* Evidence of major pulmonary vessel encasement on CT scan of the chest
* Myocardial infarction (Ml) or unstable angina in the previous 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2004-02; Primary Completion 2013-06 (Actual); Study Completion 2014-06

PRIMARY OUTCOMES:
MTID | Up to 2 years
  Defined as the dose at which =< 1 out of 6 patients experiences dose-limiting toxicity.
Systemic toxicity according to NCI Common Toxicity Criteria version 2 | Up to 6 months
PDT-related normal tissue toxicity | Up to 6 months
  Assessed by a scale with grades 0-3 being acceptable, grade 4 being unacceptable, and grade 5 being stopping study.

SECONDARY OUTCOMES:
Objective tumor response | Up to 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Samjot Dhillon, Principal Investigator — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States